CLINICAL TRIAL: NCT03351348
Title: Double Blind, Randomized, Placebo Controlled Trial of Locally Instilled Bupivacaine in the Surgical Bed After Unilateral Mastectomy Without Reconstruction
Brief Title: Bupivacaine vs Placebo for Unilateral Mastectomy Surgical Site Post-operative Pain Control
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-576
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Bupivacaine; Mastectomy; Sentinel lymph node biopsy SLNB; 17-576
MeSH Terms: conditions — Breast Neoplasms | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A prospective, double-blind, randomized, placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: Treatment assignments can be viewed only by the hospital pharmacists who are dispensing the study drugs.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline + usual post-operative medications (Active Comparator): The intervention in this study is the insertion of 20cc of saline via a drain into the mastectomy wound for 2 hours ± 30 minutes postoperatively in patients undergoing unilateral mastectomy without breast reconstruction +/- SLNB, +/- axillary dissection.
  Interventions: Behavioral: patient-reported pain scores; Other: saline
- Bupivacaine + usual post-operative medications (Experimental): The intervention in this study is the insertion of 20cc of 0.5% bupivacaine via a drain into the mastectomy wound for 2 hours ± 30 minutes postoperatively in patients undergoing unilateral mastectomy without breast reconstruction +/- SLNB, +/- axillary dissection.
  Interventions: Drug: Bupivacaine; Behavioral: patient-reported pain scores

INTERVENTIONS:
Drug: Bupivacaine — The intervention in this study is the insertion of 20cc of 0.5% bupivacaine via a drain into the mastectomy wound for 2 hours ± 30 minutes postoperatively in patients undergoing unilateral mastectomy without breast reconstruction +/- SLNB, +/- axillary dissection.
  Arms: Bupivacaine + usual post-operative medications
Behavioral: patient-reported pain scores — Will be recorded by the nurse in the PACU as per usual practice. Patients will be given a follow-up Brief Pain Inventory (short form) 6 months and 1 year after surgery to assess their level of chronic pain. Patients may be discharged when table either on the day of surgery or post-operative day 1 (on pill diary for same-day discharge patients).
Other: saline — The intervention in this study is the insertion of 20cc of saline via a drain into the mastectomy wound for 2 ± 30 minutes hours postoperatively in patients undergoing unilateral mastectomy without breast reconstruction +/- SLNB, +/- axillary dissection.
  Arms: Saline + usual post-operative medications

SUMMARY:
The purpose of this study is to compare using FDA-approved bupivacaine (a numbing medicine), along with the usual medications for post-operative pain control to using the usual medications for postoperative pain control alone. The addition of bupivacaine to the surgical wound site with the usual pain medications could better manage your pain immediately after surgery and reduce the amount of opioid medications taken after surgery. This study will allow the researchers to know whether this different approach is better, the same, or worse than the usual approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Patients undergoing unilateral mastectomy with or without SLNB or axillary dissection
* Patients scheduled for surgery at the JRSC or MSK Monmouth
* Previously enrolled patients > 6 months from contralateral mastectomy

Exclusion Criteria:

* Patients who are non-English speaking
* Patients having any immediate breast reconstructive procedure
* Patients are having bilateral mastectomy
* Patients who report a baseline pain score > 3, unrelated to a breast procedure
* Patients who take long acting opioid medication use
* Patients will be excluded if they are having their mastectomy performed with tumescence
* Patients weighing < 40kg as 20cc of bupivacaine 0.5% is greater than the maximum allowed dose
* Patients within 6 months of previous enrollment for surgery for contralateral mastectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2017-11-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
number of patients that have moderate to severe pain | up to 24 hours
  Validated measures consisting of the Comparative Pain Scale and Simplified Postoperative Nausea and Vomiting (PONV) impact scale are currently administered to postoperative patients at JRSC. The Comparative pain scale ranges from 0-10, with 0 representing no pain and 10 representing the most severe pain.
  0 = no pain 1-3 = minor pain 4-6 = moderate pain 7-10 = severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Kirstein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and follow-up only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and follow-up only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and follow-up only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and follow-up only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and follow-up only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/